CLINICAL TRIAL: NCT05216757
Title: Efficacy and Safety of Iguratimod in Patients With Hand Osteoarthritis (ESIGO) : a Randomized Control Trial
Brief Title: Efficacy and Safety of Iguratimod in Patients With Hand Osteoarthritis (ESIGO)
Acronym: ESIGO
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IGU-HOA
Record Dates: First submitted 2022-01-07; First posted 2022-01-31 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-01

CONDITIONS: Hand Osteoarthritis; Inflammatory Arthritis
Keywords: inflammatory hand osteoarthritis; iguratimod; a randomized control trial
MeSH Terms: conditions — Arthritis | interventions — iguratimod

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Iguratimod group (Active Comparator): subjects with Iguratimod
  Interventions: Drug: Iguratimod
- placebo group (Placebo Comparator): subjects with placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Iguratimod — iguratimod, 25mg bid po.
  Arms: Iguratimod group
Drug: placebo — placebo 1 tablet bid po.
  Arms: placebo group

SUMMARY:
Hand osteoarthritis is one of the most common arthritis, resulting in pain in finger and thumb base joints. The disease is characterized by pain and stiffness of the affected joints and is the most common cause of disability in aged people. Currently limited therapy options are available. Synovial inflammation is involved in the joint pain. Iguratimod is a small disease-modifying compound that can influence anti-inflammatory pathways in models of rheumatoid arthritis. It has an anabolic effect on the bone metabolism of infected joint by osteoclastogenesis inhibition and osteoblast differentiation. The investigators hypothesize that Iguratimod will alleviate pain of patient with inflammatory hand osteoarthritis, and that a beneficial effect of Iguratimod on pain will be accompanied by a decrease of synovial inflammation.

ELIGIBILITY:
Inclusion criteria

Patients to be included must meet the following criteria:

1. Age of 45-75 years.
2. Men or women.
3. Hand OA according to the ACR criteria.
4. Symptomatic interphalangeal osteoarthritis for more than 3 months (at least every other day).
5. At least 1 IPJ (DIP/PIP/IP1st) with soft tissue swelling or erythema.
6. At least 1 IPJ with positive power Doppler signal or/and synovial thickening of at least grade 2 on ultrasound.
7. Finger pain which was more than 40 mm as evaluated by visual analogue scales (VAS) (0-100 mm) in the preceding 48 hours.
8. Be able to adhere to the study visit schedule and other protocol requirements. Capable of giving informed consent and the consent must be obtained prior to any screening procedures.

Exclusion Criteria:

1. Other known medical disease that may affect joints, e.g. rheumatoid arthritis, gout, psoriatic arthritis, reactive arthritis, ankylosing spondylitis, Lyme disease, Systemic lupus erythematosus, Sjogren Syndrome, Systemic sclerosis.
2. Psoriasis.
3. involving carpometacarpal [CMC] joints, without interphalangeal joints.
4. Existence of painful syndrome of upper limbs likely to interfere with the monitoring of pain (cervicobrachial neuralgia, incapacitating carpal tunnel syndrome, joint disorders of the elbow or shoulder, poly-articular chondrocalcinosis, fibromyalgia).
5. Trigger finger, injury in joints within past 6 months.
6. Slow-acting drugs for OA (e.g. glucosamine, chondroitin, diacerhein) initiated within the previous 3 months before the study.
7. Intra-articular treatments or aspirations of any kind of any joint in the hands 3 months before screening.
8. Intra-articular corticosteroids into any joint or use of systemic corticosteroids 1 month before screening.
9. Treatment with analgesics initiated within the previous 1 month and NSAIDs initiated within the previous 2 weeks.
10. History of hand surgery within 12 months prior enrolment.
11. Participation in experimental device or experimental drug study 3 months prior to enrolment.
12. Scheduled surgery during study participation.
13. Pregnant or lactating women，planned pregnancy within the study period, 3 months after end of study treatment for female fertile participant.
14. Known blood dyscrasias and coagulation disorders.
15. Elevated alanine transaminase (AST/ALT > 2x upper normal range).
16. GRF (MDRD) < 60 mg/min/1.73m2.
17. Known viral hepatitis B or C.
18. Uncontrolled diseases, such as asthma or inflammatory bowel disease, where flares are commonly treated with oral or parenteral corticosteroids.
19. History of peptic ulcer.
20. Patients who have severe comorbidities, including cardiovascular, nervous system, pulmonary, renal, hepatic, endocrine, GI disease. Known any other condition or impairment that, in the opinion of the investigator, makes a potential participant unsuitable for participation or which obstruct participation, such as e.g. psychiatric disorders.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in patient's assessment of arthritis pain on a visual analogue scale | 12 weeks
  Change from baseline in self-reported finger joint pain previous 48 hours on a 0-100 mm scale at 12 weeks of treatment; higher value indicate worse outcome.

SECONDARY OUTCOMES:
Change from baseline in patient's assessment of arthritis pain on a visual analogue scale prior to each visit | 4 weeks, 8 weeks, 12 weeks
  Differences in self-reported finger joint pain previous 48 hours on a 0-100 mm scale at 4 weeks, 8 weeks, and 12 weeks; higher value indicate worse outcome.
Change from baseline in Australian Canadian Hand Osteoarthritis Index (AUSCAN) scores at each visit. | 4 weeks, 8 weeks, 12 weeks
  The AUSCAN Index is a self-administered questionnaire consisting of a 15-item scale which measures pain (5 items), stiffness (1 item) and degree of disability/physical function (9 items) during the preceding 48 hours; higher value indicate worse outcome.
Change from baseline in Functional Index for Hand Osteoarthritis (FIHOA) | 12 weeks
  The Functional Index for Hand Osteoarthritis (FIHOA) is a leading assessment tool for hand OA-related functional impairment; higher value indicate worse outcome.
Change from baseline in Health Assessment Questionnaire Disability Index (HAQ) | 12 weeks
  Change from baseline in Health Assessment Questionnaire Disability Index (HAQ) at week 12; higher value indicate worse outcome.
Change from baseline in the Scores of SF-36 questionnaire | 12 weeks
  Change from baseline in SF-36, including physical and mental component sores (PCS and MCS) at week 12; higher value indicate worse outcome.
Change from baseline in Michigan Hand Outcomes Questionnaire (MHOQ) | 12 weeks
  Michigan Hand Outcomes Questionnaire (MHOQ) pain and physical function subscales; function subscale range 10-50, higher value indicate worse outcome; task subscale range 17-85, higher value indicate worse outcome; work subscale range 5-25, higher value indicate worse outcome; pain subscale range 10-48, higher value indicate better outcome.
Change from baseline in Ultrasound record | 12 weeks
  Ultrasound record: number of finger joints with synovial thickening and power Doppler signals.
Change from baseline in OMERACT hand OA magnetic resonance imaging score | 12 weeks
  OMERACT hand OA magnetic resonance imaging score includes synovitis (0-3), erosive damage(0-3), cyst (0-3), osteophyte (0-3), cartilage space loss(0-3), malalignment (0-3), and bone marrow lesions (0-3); higher value indicate worse outcome

OTHER OUTCOMES:
Change from baseline in Erythrocyte Sedimentation Rate (ESR) | 12 weeks
  Erythrocyte Sedimentation Rate (ESR); higher value indicate worse outcome.
Change from baseline in C Reactive Protein (CRP) | 12 weeks
  C Reactive Protein (CRP); higher value indicate worse outcome.
Change from baseline in patient's global assessment of disease activity on a visual analogue scale | 12 weeks
  Change from baseline in patient's global assessment of disease activity previous 48 hours on a 0-100 mm scale at 12 weeks of treatment; higher value indicate worse outcome.
Change from baseline of physician's global assessment of disease activity on a visual analogue scale | 12 weeks
  Change from baseline in physician's global assessment of disease activity previous 48 hours on a 0-100 mm scale at 12 weeks of treatment; higher value indicate worse outcome.
Change from baseline in Fingertip-to-palm distance | 12 weeks
  Change from baseline in Fingertip-to-palm distance, cm
Change from baseline in grip strength | 12 weeks
  Change from baseline in grip strength, kg
Swelling and Tender joint count, assessed by physician joint count | 12 weeks
  Swelling and Tender joint count, assessed by physician joint count